CLINICAL TRIAL: NCT01594918
Title: A Phase I Study of Cabazitaxel, Mitoxantrone, and Prednisone (CAMP) for Patients With Metastatic Castration-Resistant Prostate Cancer and no Prior Chemotherapy
Brief Title: Phase I Cabazitaxel, Mitoxantrone, and Prednisone Metastatic Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rahul Aggarwal (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor-Investigator, Rahul Aggarwal, Assistant Clinical Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCSF Protocol No. 11951
Record Dates: First submitted 2012-05-07; First posted 2012-05-09 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: metastatic; CRPC; prostate; CAMP
MeSH Terms: conditions — Neoplasm Metastasis | interventions — cabazitaxel; XRP6258; Mitoxantrone; Prednisone; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cabazitaxel, Mitoxantrone, Prednisone (Experimental)
  Interventions: Drug: Cabazitaxel; Drug: Mitoxantrone; Drug: Prednisone; Drug: Pegfilgrastim

INTERVENTIONS:
Drug: Cabazitaxel — 25 mg/m2 or 20 mg/m2, IV, once every 21 days
  Other Names: Jevtana®; XRP6258; RPR116258
Drug: Mitoxantrone — 4 mg/m2, 6 mg/m2, 8 mg/m2, 10 mg/m2, or 12 mg/m2, IV, once every 21 days
  Other Names: Novantrone
Drug: Prednisone — 5 mg PO BID
Drug: Pegfilgrastim — 6 mg, SC, once every 21 days
  Other Names: Neulasta

SUMMARY:
The purpose of this study is to test the safety of cabazitaxel, mitoxantrone, and prednisone (CAMP) in combination at different dose levels and to determine the highest dose that does not cause bad side effects. The investigators want to find out what effects, good and/or bad, CAMP has on patients and their metastatic castration-resistant prostate cancer.

DETAILED DESCRIPTION:
This is a Phase I, open label, dose-finding, multicenter clinical trial to establish the maximum tolerated dose (MTD) and dose limiting toxicities (DLT) of cabazitaxel (25 mg/m2 IV q21 days) in combination with mitoxantrone (4-12 mg/m2 IV q21 days) and prednisone (5mg orally BID) in patients with metastatic CRPC who have not undergone prior chemotherapy for metastatic disease.

Up to five cohorts will be enrolled to determine the MTD and DLT profile of this combination. An accelerated titration design method is being used in order to minimize the number of patients exposed to subtherapeutic doses of mitoxantrone.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the prostate.

2. Progressive metastatic prostate cancer (positive bone scan or measurable disease) despite castrate levels of testosterone (either from orchiectomy or LHRH agonist therapy).

3. Patients may have either non-measurable disease OR measurable disease

4. All patients must have a PSA ≥ 2 ng/mL.

5. Progressive disease based on any one of the following:

1. transaxial imaging
2. a rise in PSA
3. radionuclide bone scan

   Patients whose sole manifestation of progression is an increase in disease-related symptoms are not eligible.
   1. For patients with measurable disease, progression will be defined by the RECIST criteria.
   2. For patients with non-measurable disease, a positive bone scan and elevated PSA will be required. PSA evidence for progressive prostate cancer during or after first-line chemotherapy consists of a PSA level of at least 2 ng/ml which has risen on at least 2 successive occasions, at least one week apart. If the confirmatory PSA (#3) value is less (i.e., #3b) than the screening PSA (#2) value, then an additional test for rising PSA (#4) will be required to document progression for the purposes of eligibility.
   3. Radionuclide bone scan: new metastatic lesions

      6. Testosterone < 50 ng/dL. Patients must continue primary androgen deprivation with an LHRH analogue if they have not undergone orchiectomy.

      7. ECOG Performance Status 0 -2.

      8. Required Laboratory values:

   <!-- -->

   1. Creatinine < 1.5 x upper limits of normal (ULN). If Cr. > 1.5 x ULN, then calculated creatinine clearance > 40cc/min.
   2. ALT and AST within normal limits
   3. Absolute neutrophil count > 2,000/mm3
   4. Platelets > 100,000/ mm3
   5. Hemoglobin > 8.0 gm/dL
   6. Total bilirubin within normal limits

      9. Ejection fraction by MUGA scan or echocardiogram ≥ lower limit of institutional normal.

      10. Patients receiving hormonal therapy (i.e. any dose of megestrol acetate (Megace), Proscar (finasteride), any herbal product known to decrease PSA levels (e.g., Saw Palmetto and PC-SPES) other than LHRH agonist/antagonist or a stable dose of corticosteroid from a prior chemotherapy regimen must discontinue the agent for at least 4 weeks prior to enrollment. Progressive disease must be documented after discontinuation of the hormonal therapy.

      11. No other systemic therapies for prostate cancer within 28 days prior to initiation of this protocol.

      12. Prior radiation therapy completed ≥ 4 weeks prior to enrollment.

      13. No history of radiopharmaceuticals (strontium, samarium) for prostate cancer treatment.

      14. Patients must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry, for the duration of study participation and for 3 months after discontinuing therapy. Should a patient's sexual partner become pregnant or suspect she is pregnant while the patient is participating in this study, he should inform the treating physician immediately.

      15. Life expectancy > 12 weeks.

      16. Age ≥ 18 years

      17. Inclusion of Minorities: Men and members of all ethnic groups are eligible for this trial.

      Exclusion Criteria:
      1. Patients with significant cardiovascular disease including congestive heart failure (NYHA class III or IV), active angina pectoris or myocardial infarction within 6 months.
      2. Patients with serious intercurrent infections, or nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the complications of this therapy.
      3. Patients with psychiatric illness/social situations that would limit compliance with study requirements.
      4. Patients with pre-existing neuropathy greater than CTCAE Grade 1 (motor or sensory).
      5. Patients with known prior severe hypersensitivity reactions to cabazitaxel or other agents containing polysorbate 80.
      6. Patients with known active brain metastases are excluded because of their poor prognosis. Head CT is NOT routinely required prior to enrollment. Patients with treated, asymptomatic brain metastasis will be eligible for enrollment.
      7. Patients with a "currently active" second malignancy other than non-melanoma skin cancer are excluded. [Patients are not considered to have a "currently active" malignancy if they have completed therapy and are considered by their physician to be at less than 30% risk of relapse.]
      8. Concurrent use of moderate to strong CYP3A4 inhibitors is not allowed.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-06; Primary Completion 2016-08 (Actual); Study Completion 2017-06-23 (Actual)

PRIMARY OUTCOMES:
Determination of the maximum tolerated dose (MTD) of the combination of cabazitaxel and mitoxantrone/prednisone as chemotherapy for patients with metastatic CRPC who have not received prior chemotherapy for metastatic disease. | Participants will be followed for the duration of treatment, an expected average of 4 months.

SECONDARY OUTCOMES:
Dose Limiting Toxicity (DLT) | Participants will have AE/Toxicity evaluations every 21 days. Average study participation is approximately 4 months.
  Number of Grade 3 or greater non-hematologic toxicity recorded.
Reduction in Prostate Specific Antigen (PSA), of the combination of cabazitaxel and mitoxantrone/prednisone in patients with metastatic CRPC who have not received prior chemotherapy for metastatic disease. | Participants will have PSA assessments every 21 days. Average study participation is approximately 4 months.
Efficacy of drug combination including objective response rate and duration of response | Participants will be followed for the duration of treatment, an expected average of 4 months.

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Aggarwal, MD, Study Chair — University of California, San Francisco
Locations (3):
- United States (3):
  - Mayo Clinic, Scottsdale, Arizona
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee